CLINICAL TRIAL: NCT00282126
Title: Potassium Citrate to Prevent Age Related Bone Loss: Pilot Study
Brief Title: Potassium Citrate to Prevent Age Related Bone Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: N01 AR052275; 27653
Record Dates: First submitted 2006-01-23; First posted 2006-01-25 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Osteoporosis
Keywords: Calcium balance
MeSH Terms: conditions — Osteoporosis | interventions — Potassium Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Participants will receive 90 meq of potassium citrate.
  Interventions: Dietary Supplement: Potassium citrate
- 2 (Experimental): Participants will receive 60 meq of potassium citrate.
  Interventions: Dietary Supplement: Potassium citrate
- 3 (Placebo Comparator): Participants will receive placebo.
  Interventions: Dietary Supplement: Potassium citrate

INTERVENTIONS:
Dietary Supplement: Potassium citrate — kcitrate

SUMMARY:
Osteoporosis, a disease in which the bones become weak and are more likely to break, is a major health problem in the United States. Too much acid in the body appears to be linked to loss of calcium via urine, bone loss, and muscle breakdown. The purpose of this study is to determine the effect of various doses of potassium citrate, a supplement that can neutralize acid, on bone density and muscle mass in older, healthy adults.

DETAILED DESCRIPTION:
Over 10 million adults in the United States have osteoporosis, and another 18 million have low bone mass, a risk factor for developing this disease. Each year, approximately 1.5 million fractures are associated with osteoporosis. Adequate intake of calcium and vitamin D is the current nutritional approach to preventing age-related bone loss. However, even with sufficient levels of these nutrients, bone loss can still occur. Too much acid in the body, caused by diet, aging, and protein metabolism, appears to be linked to loss of calcium via urine, bone loss, and muscle breakdown. Potassium citrate can neutralize acids. The purpose of this study is to determine the effect of various doses of potassium citrate on bone density and muscle mass in older, healthy adults.

This study will last 6 months. Baseline measurements will take place from Weeks 1 through 4. During this time, participants will first receive a placebo over a 2-week period. Participants will then undergo a calcium balance study, involving consumption of certain study foods for 12 days and an overnight stay at the research unit for a calcium absorption test. The calcium balance study will be followed by blood collection. At Week 5, participants will be randomly assigned to receive either potassium citrate or placebo daily. For the first 9 weeks of treatment, there will be weekly blood collection and periodic urine collection for all participants. At Month 6, blood and urine will again be collected, and participants will complete questionnaires on diet and physical activity, and a second calcium balance study.

ELIGIBILITY:
Inclusion Criteria:

* Good general health

Exclusion Criteria:

* Abnormal kidney, liver, or bone function
* Currently taking medications that might affect potassium or bone

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-01; Primary Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
calcium balance | six months

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Sellmeyer, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States